CLINICAL TRIAL: NCT00844506
Title: p53 Synthetic Long Peptides Vaccine With Cyclophosphamide for Ovarian Cancer a Phase II Trial
Brief Title: p53 Synthetic Long Peptides Vaccine With Cyclophosphamide for Ovarian Cancer
Acronym: ISA-P53-CTX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ISA Pharmaceuticals B.V. (Industry); Dutch Cancer Society (Other)
Responsible Party: Prof. Dr. H.W. Nijman, University Medical Centre Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISA-P53-CTX; EUDRACT 2007-007734-19; CCMO NL21308.000.07
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer patients with recurrent disease
MeSH Terms: conditions — Ovarian Neoplasms | interventions — p53 synthetic long peptide vaccine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: P53-SLP vaccine — The P53-SLP vaccine is a vaccine consisting of a total of 10 long (30 amino acids on average length) peptides, covering the p53 protein sequence from amino acid 70 to 251, combined with Montanide ISA51 an adjuvant with a sustained dendritic cell activating ability. Patients will be immunised subcutaneously with the peptide vaccine four times with a three week interval (300μg/peptide).
Drug: Cyclophosphamide — Two days prior to each peptide vaccination, patients will receive 300mg/m2 cyclophosphamide i.v.
  Other Names: Endoxan; Cytoxan

SUMMARY:
The purpose of this study is to determine whether the addition of cyclophosphamide to the treatment with the p53-SLP vaccine improves clinical efficacy and immunogenicity of the p53-SLP vaccine in ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histological proven epithelial ovarian carcinoma.
* At least 4 weeks after termination of the last course of chemotherapy.
* Rising CA-125 serum levels after "first line" treatment and no measurable disease according to the RECIST (Response Evaluation Criteria in Solid Tumours) criteria, or Rising CA-125 serum levels after "first line" treatment with measurable disease according to the RECIST (Response Evaluation Criteria in Solid Tumours) criteria, but not willing or otherwise not fit to receive "second line" chemotherapy.
* Age 18 years or older, and an life expectancy of at least 3 months.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Performance status 0 to 2 (WHO scale).
* Adequate hepatic, renal, and bone marrow function as defined:

ASAT < 100 U/l; ALAT < 113 U/l; PT 9-12 seconds; APTT 23-33 seconds; creatinine < 135 μmol/l; WBC > 3.0 x 109/L; platelets > 100 x 109/L; hemoglobin > 6.0 mmol/l.

- Adequate venous access for blood collection and i.v. administration of cyclophosphamide.

Exclusion Criteria:

* Pregnancy and / or breast feeding.
* (A)symptomatic cystitis.
* Other malignancies (previous or current), except basal or squamous cell carcinoma of the skin.
* Immunosuppressive agents, except for topical and inhalation corticosteroids.
* Prior therapy with a biological response modifier.
* Any other major disease that may interfere with the conduct of the study (e.g. uncontrolled hypertension, severe and/or unstable heart disease, neurological and psychiatric disorders).
* Signs or symptoms of CNS metastases.
* Known substance abuse (drug or alcohol).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Clinical responses to the p53 synthetic long peptide vaccine preceded by cyclophosphamide will be assessed by measurement of serum CA-125 levels and CT-scan. | day 105 - 126 after first gift of cyclophosphamide
Immunogenicity will be evaluated by assessing induction and frequency of p53-specific T cells by proliferation and IFN-γ ELISPOT. | after fourth immunization

SECONDARY OUTCOMES:
Safety of the vaccine preceded by cyclophosphamide will be assessed by monitoring the incidence and severity of adverse events using Common Terminology Criteria for Adverse Events v3.0. | durante study

CONTACTS AND LOCATIONS:
Overall Officials: H. W. Nijman, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Speetjens FM, Kuppen PJ, Welters MJ, Essahsah F, Voet van den Brink AM, Lantrua MG, Valentijn AR, Oostendorp J, Fathers LM, Nijman HW, Drijfhout JW, van de Velde CJ, Melief CJ, van der Burg SH. Induction of p53-specific immunity by a p53 synthetic long peptide vaccine in patients treated for metastatic colorectal cancer. Clin Cancer Res. 2009 Feb 1;15(3):1086-95. doi: 10.1158/1078-0432.CCR-08-2227. PMID 19188184
- [Background] Lambeck A, Leffers N, Hoogeboom BN, Sluiter W, Hamming I, Klip H, ten Hoor K, Esajas M, van Oven M, Drijfhout JW, Platteel I, Offringa R, Hollema H, Melief K, van der Burg S, van der Zee A, Daemen T, Nijman H. P53-specific T cell responses in patients with malignant and benign ovarian tumors: implications for p53 based immunotherapy. Int J Cancer. 2007 Aug 1;121(3):606-14. doi: 10.1002/ijc.22710. PMID 17415711